## Kidney Transplants in Hepatitis C Negative Recipients With Hepatitis C Viremic Donors

NCT04575896

**September 29, 2020** 



Principal Investigator: Niraj Desai, MD Application No.: IRB00237097

> If appropriate for this study, a scanned copy of the signed consent form should be uploaded to

the participant's Epic/EMR record.

Patient I.D. plate

# RESEARCH PARTICIPANT INFORMED CONSENT AND PRIVACY AUTHORIZATION FORM

Protocol Title: Kidney transplants in hepatitis C negative recipients with

hepatitis C viremic donors. An open-label, non-randomized pilot study to determine the safety and efficacy of two weeks of fixed-dose glecaprevir and pibrentasvir as pre- and post-exposure

prophylactic therapy.

**Application No.:** IRB00237097

**Supported By:** The Johns Hopkins Department of Surgery

Principal Investigator: Niraj Desai, MD

**Assistant Professor of Surgery** 

720 Rutland Ave., Ross Building Room 765

Baltimore, MD 21205 Phone: 410-614-8297 Fax: 410-367-2396

You are being asked to join a research study. Participation in this study is voluntary. Please read this consent form carefully and take your time making your decision. Even if you decide to join now, you can change your mind later.

## 1. Research Summary (Key Information):

The information in this section is intended to be an introduction to the study only. Complete details of the study are listed in the sections below. If you are considering participation in the study, the entire document should be discussed with you before you make your final decision. You can ask questions about the study now and at any time in the future.

The purpose of this research is to determine if giving an investigational study drug combination called Glecaprevir/Pibrentasvir (G/P) for 2 weeks is safe and effective in preventing the HCV virus (hepatitis C virus) from infecting a kidney transplant recipient when a kidney from a kidney donor with the virus is used for transplant.

G/P belongs to a group of medications called direct-acting antiviral agents (DAAs). These drugs are intended to prevent the Hepatitis C Virus from multiplying and spreading in the human body.



Principal Investigator: Niraj Desai, MD Application No.: IRB00237097

Approximately 10 subjects who are on the deceased donor kidney waiting list are expected to participate in this study at Johns Hopkins. If you decide to be in this study and are eligible, your participation will last up to 14 weeks. This includes a 2-week study drug administration period and a 12-week follow-up period. There are risks to the drug that are described later in this document. Some risks could be serious and not all of the side effects/risks are known.

You may or may not benefit directly from being in the study and there is no payment for participation.

## 2. Why is this research being done?

This research is being done to determine if giving an investigational study drug combination called Glecaprevir/Pibrentasvir (G/P) for 2 weeks is safe and effective in preventing the HCV virus from infecting a kidney transplant recipient when a kidney from a kidney donor with the HCV is used for transplant.

G/P belongs to a group of medications called direct-acting antiviral agents (DAAs). These drugs are intended to prevent the Hepatitis C Virus from multiplying and spreading in the human body.

Glecaprevir/Pibrentasvir are already approved and used for 8 weeks to treat HCV infection. The use of Glecaprevir/Pibrentasvir for 2 weeks in preventing HCV infection is investigational. The word "investigational" means that Glecaprevir/Pibrentasvir are not approved for marketing by the Food and Drug Administration (FDA) and are still being tested. The FDA is allowing for Glecaprevir/Pibrentasvir to be used in this study.

## Who can join this study?

People who are 18 years or older, who are on the deceased donor kidney waiting list at Johns Hopkins Hospital awaiting their first or second kidney for transplant, and who have no available living donors may join.

## How many people will be in this study?

We will enroll 10 people in this study.

## 3. What will happen if you join this study?

If you agree to be in this study, we will ask you to do the following things:

#### **Screening phase:**

Patients who are waiting for a kidney transplant at Johns Hopkins Hospital and meet the above criteria will be approached with this informed consent form and screened for enrollment in the study. Your medical record will be closely reviewed and your blood may be drawn. We will also review the medications you are currently taking to see if any of them should not be given with the study drug. If you are currently taking one of these medications and it cannot be safely discontinued or substituted with another medication you will not be able to continue to participate in the study and you will not be listed with a status of "willing to accept an HCV+ organ". If you are prescribed any new medications after signing this consent, it is important that you report it to the study doctor at the time it is prescribed.

#### **Donor Identification:**

Once you provide informed consent for this study, and it has been confirmed that your medications are safe to give with the study drug, you will be listed in the United Network for Organ Sharing (UNOS) with a status of "willing to accept an HCV+ organ". The Johns Hopkins transplant team will then receive HCV+ donor kidney offers for participants of this study. If an HCV+ donor is identified who meets the requirements of this study, you will be offered the organ. If you accept, you will become an active study participant.



Principal Investigator: Niraj Desai, MD Application No.: IRB00237097

## Active phase, transplant and study drug regimen:

After you have signed consent and prior to you receiving a transplant we will draw approximately 9 tablespoons of blood so we can measure how your immune system responds to getting a hepatitis C infected organ. If your transplant does not occur within 12 months of this blood being drawn, we may need to repeat the blood draw. At the time of your admission to the hospital for your transplant, you will undergo the standard pre-operative preparation, including laboratory testing, chest X-ray, electrocardiogram (EKG), and urine analysis. In addition, a blood sample for this study will be drawn. Your initial dose of glecaprevir and pibrentasvir will be administered by your nurse when you are called to the operating room.

Except for the study drug, your kidney transplant and postoperative care will be the same as for patients not on this study. After your transplant, you will be given glecaprevir and pibrentasvir every day. Most kidney transplant recipients are able to take medicine by mouth within eight hours after their transplant.

Discharge from the hospital is typically between 7 and 10 days after the transplant, once your new kidney is functioning properly, you are tolerating a regular diet, and you have normal bowel and bladder function. During your hospitalization, we will discuss your medications, including glecaprevir and pibrentasvir, and planned follow-up visits several times.

The study drug regimen phase of the study will be 2 weeks; we will monitor you closely for HCV. These drugs have been shown to be effective in preventing HCV complications. However, if the virus does become detectable, we will treat your hepatitis C according to the most current clinical standard.

## Follow-up:

You will have study visits 1, 2, 4, and 12 weeks after you stop taking the study drugs. During study visits, we will review your medical record, complete a physical exam, and take a blood sample for the study. We may also ask you to come in for a visit 24 weeks after you stop taking the study drugs based on the results from your week 12 bloodwork.

## Will research test results be shared with vou?

This study may involve research tests that may produce information that could be useful for your clinical care. Information about your study participation will be included in your medical record and we will share this information with you.

## How long will you be in the study?

You will be in this study for at least 14 weeks after your kidney transplant. However, we will continue to collect information about your health for at least 12 months after your transplant.

## 4. What happens to data and biospecimens that are collected in the study?

Johns Hopkins and our research partners work to advance science and public health. The data and biospecimens we collect from you are important to this effort.

Biospecimens may include any of the following: blood, tissue, saliva, urine, bone marrow, cells, etc. Most biospecimens contain DNA, which is the genetic code for each person.

If you join this study, you will not own the data and/or biospecimens collected from you as part of this research study. If researchers use them to create a new product or idea, including those that may have commercial value, you will not benefit financially from these efforts.



Principal Investigator: Niraj Desai, MD Application No.: IRB00237097

## What testing or procedures may be done with your biospecimens?

Your biospecimens may be used for a variety of research purposes. The specific testing that is included in this study is taking blood samples to test for HCV plasma RNA levels and measurement of T cell responses to HCV peptides. Allograft biopsies will be performed if there is concern for rejection or other causes of graft dysfunction.

## How will your data and/or biospecimens be shared now and in the future?

Sharing data and/or biospecimens is part of research and may increase what we can learn from this study.

Often, data/biospecimen sharing is required as a condition of funding or for publishing study results. It also is needed to allow other researchers to validate study findings and to come up with new ideas.

Your data and/or biospecimens may be shared:

- directly with research collaborators, other researchers, sponsors, government agencies, publishers of papers and other research partners
- through government or other databases/repositories

Data/biospecimen sharing could change over time, and may continue after the study ends.

We will do our best to protect and maintain your data/biospecimens in a safe way. Generally, if we share your data/biospecimens without identifiers (such as your name, address, and date of birth) further review and approval by an IRB is not needed. However, when we share data/biospecimens, we limit the uses of the information and whether these data/biospecimens can be shared with another research team. If data/biospecimens are shared with identifiers, further IRB review and approval may be needed and the IRB will determine whether additional consent is required.

Johns Hopkins researchers may also use the biospecimens collected in this study for future research purposes, which may include gene sequencing and genetic testing. Each cell contains your complete DNA. Gene sequencing of your DNA provides researchers with the code to your genetic material. This future research may be unrelated to the current study and may include outside collaborators.

Because science constantly advances, we do not yet know what future testing may include. If biospecimens are tested/used in ways not described above, further IRB review and approval may be needed and the IRB will determine whether additional consent is required.

If you are not comfortable with the use of your data/biospecimens in future research, you may not want to participate in this study.

## 5. What are the risks or discomforts of the study? Risks of Glecaprevir and Pibrentasvir

The most common side effects with these study drugs are headache, tiredness, nausea, and diarrhea. In rare cases, there were bilirubin elevations that decreased upon completing the drug.

There is a very rare possibility of acquiring hepatitis C, which may result in fulminant (sudden and rapidly progressing) hepatitis and death. If you develop hepatitis, the study will not be responsible for the cost of your treatment.



Principal Investigator: Niraj Desai, MD

Application No.: IRB00237097

#### **Blood Draw**

Taking blood may cause discomfort, bleeding, or bruising where the needle enters the body. In rare cases, it may result in fainting. There is a small risk of infection.

## **Identifiable private information**

There is the risk that information about you may become known to people outside this study. To protect against this, the study information will be kept in password protected computers in locked rooms that are accessible only to study staff.

## Unknown risk

There may be side effects and discomforts that are not yet known.

#### **6.** Are there risks related to pregnancy?

To date there is no adequate human data available to establish whether or not the study drug poses a risk to an embryo or fetus.

For female participants, extreme care must be taken to avoid pregnancy during this study and for up to 6 months after the last dose of glecaprevir and pibrentasvir. For male participants, extreme care must be taken to avoid pregnancy in female partners during this study and for up to 6 months following completion of the study regimen. If you are pregnant, intending to become pregnant, or currently nursing (breastfeeding) a child, you cannot be in this study. If you are a man whose partner is currently pregnant or wishing to become pregnant, you cannot be in this study.

You must protect yourself or your partner from becoming pregnant before, during, and after the study. Women, and men with female partners capable of becoming pregnant, must use effective methods of birth control as described below. Your study doctor will need to document what type(s) of birth control you are using.

#### Women only:

Women who can get pregnant should not take study drug(s) unless they and their partner do not have intercourse ever or are using 2 methods of birth control for the duration of the study (starting 3 weeks prior to the Day 1 visit) and for a minimum of 6 months after last dose of study drug or longer as directed by your study doctor.

At least one method of birth control must be a condom used correctly by your male partner. Your study doctor will discuss with you other methods of birth control that can be used in combination with a condom.

Women who can get pregnant must have a negative pregnancy test at time of admission for transplant, and prior to taking the first dose of study drug.

You must tell your study doctor immediately if you become pregnant while in this study and for 6 months after stopping the study drug, or for as long as you have been directed by your study doctor to use contraception. The study doctor will tell you about the possible risks to the embryo or fetus and options available to you.

In the event of a positive urine pregnancy result, you will be instructed to return to the study clinic as soon as possible for a serum (blood) pregnancy test.



Principal Investigator: Niraj Desai, MD Application No.: IRB00237097

Men only:

If you have a female partner who cannot become pregnant, you must still consistently and correctly use a condom.

If you have a female partner who can become pregnant, you and your partner must use two forms of birth control for the entire study and for a minimum of 6 months after the last dose of study drug. You must use a condom while your female partner uses 1 other method of birth control. Your study doctor will discuss with you other methods of birth control that can be used in combination with a condom.

If your female sex partner becomes pregnant while you are in the study or within 6 months after your last dose of study drug, it is unknown if the study drug will do harm to an embryo or fetus. If you have a female partner who becomes pregnant or suspects that she has become pregnant while you are in the study or within 6 months after your last dose of study drug, you will be required to notify your study doctor immediately.

As the risks to your partner and the embryo or fetus are not known, it is recommended for your partner to receive appropriate prenatal care. Your study doctor may need to disclose to your partner details of this study and your taking part in it.

Male participants must also agree not to donate sperm from the time you first take your first dose of study drug until 6 months after the last dose of study drug

Please note: Hormonal birth control may be more effective when taken for at least 3 months. Even if you and your female partner use a medically proven birth control method, you could still cause your partner to become pregnant.

Please share this information with your partner.

## 7. Are there benefits to being in the study?

You may or may not directly benefit from this study. In some cases patients that are willing to accept an organ from an HCV-infected donor will receive an organ offer sooner than if they were not willing to accept. This may or may not have a survival benefit to being on or staying on dialysis. If you take part in this study, you may help others in the future.

## 8. What are your options if you do not want to be in the study?

You may or may not directly benefit from this study. In some cases patients that are willing to accept an organ from an HCV-infected donor will receive an organ offer sooner than if they were not willing to accept. This may or may not have a survival benefit to being on or staying on dialysis. If you take part in this study, you may help others in the future.

You do not have to join this study. Other options include waiting for an organ from a non-infected donor. If you do not join, your care at Johns Hopkins will not be affected.

## 9. Will it cost you anything to be in this study?

You will receive a separate Insurance and Research Participant Financial Responsibility Information Sheet.

This Sheet will give you the following information:



Principal Investigator: Niraj Desai, MD Application No.: IRB00237097

• The procedures, tests, drugs or devices that are part of this research and that will be paid for by the study (no cost to you).

• The procedures, tests, drugs or devices that will be billed to you and/or your health insurer. If you have health insurance, you will be responsible for any co-pays or deductibles not covered by your insurance.

## 10. Will you be paid if you join this study?

No. However, you will receive a parking pass at time of transplant and each post-transplant study visit.

## 11. Can you leave the study early?

- You can agree to be in the study now and change your mind later.
- If you wish to stop, please tell us right away.
- Leaving this study early will not stop you from getting regular medical care.

•

If you leave the study early, Johns Hopkins may use or share your health information that it has already collected if the information is needed for this study or any follow-up activities.

## 12. Why might we take you out of the study early?

You may be taken out of the study if:

- Staying in the study would be harmful.
- You need treatment not allowed in the study.
- You fail to follow instructions.
- You become pregnant.
- The study is cancelled.
- There may be other reasons to take you out of the study that we do not know at this time.

If you are taken out of the study early, Johns Hopkins may use or give out your health information that it has already collected if the information is needed for this study or any follow-up activities.

# 13. How will your privacy be maintained and how will the confidentiality of your data be protected?

#### HIPAA Authorization for Disclosure of Protected Health Information

## What information is being collected, used, or shared?

To do this research, we will need to collect, use, and share your private health information. By signing this document, you agree that your health care providers (including both Johns Hopkins Medicine and others) may release your private health information to us, and that we may use any and all of your information that the study team believes it needs to conduct the study. Your private information may include things learned from the procedures described in this consent form, as well as information from your medical record (which may include information such as HIV status, drug, alcohol or STD treatment, genetic test results, or mental health treatment).

## Who will see, use or share the information?

The people who may request, receive, or use your private health information include the researchers and their staff. Additionally, we may share your information with other people at Johns Hopkins, for example if needed for your clinical care or study oversight. To improve coordination of your research and clinical care, some information about the study you join will be included in your electronic medical record.



Principal Investigator: Niraj Desai, MD Application No.: IRB00237097

By signing this form, you give permission to the research team to share your information with others outside of Johns Hopkins. This may include the sponsor of the study and its agents or contractors, outside providers, study safety monitors, government agencies, other sites in the study, data managers and other agents and contractors used by the study team.

We try to make sure that everyone who sees your information keeps it confidential, but we cannot guarantee that your information will not be shared with others. If your information is disclosed by your health care providers or the research team to others, federal and state confidentiality laws may no longer protect it.

## Do you have to sign this Authorization?

You do not have to sign this Authorization, but if you do not, you may not join the study.

## How long will your information be used or shared?

Your Authorization for the collection, use, and sharing of your information does not expire. Additionally, you agree that your information may be used for similar or related future research studies.

## What if you change your mind?

You may change your mind and cancel this Authorization at any time. If you cancel, you must contact the Principal Investigator in writing to let them know by using the contact information provided in this consent form. Your cancellation will not affect information already collected in the study, or information that has already been shared with others before you cancelled your authorization.

## How will your information be protected?

There is the risk that information about you may become known to people outside this study. To protect against this, all samples will be stored using a de-identified label that does not contain personal identifiers. Any collected data will also be de-identified and labeled with a code and the key to the code will be kept in a password-protected computer at Johns Hopkins that will only be accessible to the study's investigators and research staff.

#### **14.** Will the study require any of your other health care providers to share your health information with the researchers of this study?

As a part of this study, the researchers may ask to see your health care records from your other health care providers. You will be asked to give us a list of other health care providers that you use.

#### 15. What treatment costs will be paid if you are injured in this study?

Johns Hopkins does not have a program to pay you if you are hurt or have other bad results from being in the study. However, medical care at Johns Hopkins is open to you as it is to all sick or injured people.

The costs for any treatment or hospital care you receive as the result of a study-related injury that are not covered by a health insurer will be billed to you.

By signing this form, you will not give up any rights you have to seek compensation for injury.

#### 16. What other things should you know about this research study?

During the study, we will tell you if we learn any new information that might affect whether you wish to continue to participate.



Principal Investigator: Niraj Desai, MD Application No.: IRB00237097

A description of this clinical trial will be available on http://www.ClinicalTrials.gov, as required by U.S. Law. This Web site will not include information that can identify you. At most, the Web site will include a summary of the results. You can search this Web site at any time. If you would like to review the information for this study, or a summary of the results, ask the study team doctor for the ClinicalTrials.gov study registration number.

## What is the Institutional Review Board (IRB) and how does it protect you?

This study has been reviewed by an Institutional Review Board (IRB), a group of people that reviews human research studies. The IRB can help you if you have questions about your rights as a research participant or if you have other questions, concerns or complaints about this research study. You may contact the IRB at 410-502-2092 or jhmeirb@jhmi.edu.

## What should you do if you have questions about the study, or are injured or ill as a result of being in this study?

Call the principal investigator, Dr. Niraj Desai at 410-614-8297. If you wish, you may contact the principal investigator by letter. The address is on page one of this consent form. If you cannot reach the principal investigator or wish to talk to someone else, call the IRB office at 410-502-2092.

If you have an urgent medical problem or think you are injured or ill because of this study, call 911 or go to your local emergency department. You should also call Dr. Niraj Desai at 410-614-8297 during regular office hours and at 314-392-7743 after hours and on weekends. If this doctor is not available, the operator will page the "on call physician."

## 17. Optional Study Components:

This part of the consent form is about optional component(s) of the study that you can choose to take part in or not. You can still take part in the main study even if you say "no" to this/these optional component(s).

#### **Future Contact**

We would like your permission for our research team to contact you in the future. Please note that your decision below does not prevent other researchers at Johns Hopkins from contacting you about other research.

| Please sign and date your choice below: | | |
|-----------------------------------------|--------------------------|------|
| YES [ | | |
| | Signature of Participant | Date |
| No□ | i <u></u> | |
| | Signature of Participant | Date |

Principal Investigator: Niraj Desai, MD Application No.: IRB00237097

## 18. What does your signature on this consent form mean?

Your signature on this form means that you have reviewed the information in this form, you have had a chance to ask questions, and you agree to join the study. You will not give up any legal rights by signing this consent form.

## WE WILL GIVE YOU A COPY OF THIS SIGNED AND DATED CONSENT FORM

| Signature of Participant | (Print Name) | Date/Time |
|---|---|---|
| Signature of Person Obtaining Consent | (Print Name) | Date/Time |
| digitative of Ferson Comming Consent | (Time Nume) | Bute, Time |
| | (D: 1) | D (T) |
| Signature of Interpreter/Witness to Consent Procedures | (Print Name) | Date/Time |
| (Required for studies enrolling non-English speakers using the shor | t form process or otherwise as determined r | equired by the IRB) |
| I have received the separate Insurance and Research Par | ticinant Financial Pasnansihility Info | ormation Shoot |
| i have received the separate insurance and Research i ar | ticipant Financial Responsibility fine | mation Sheet. |
| Signature of Participant, LAR or Parent/Guardian | (Print Name) | Date/Time |

NOTE: A COPY OF THE SIGNED, DATED CONSENT FORM MUST BE KEPT BY THE PRINCIPAL INVESTIGATOR AND A COPY MUST BE GIVEN TO THE PARTICIPANT. IF APPROPRIATE FOR THIS STUDY, A SCANNED COPY OF THE SIGNED CONSENT FORM SHOULD BE UPLOADED TO THE PARTICIPANT'S EPIC/EMR RECORD (UNLESS NO MEDICAL RECORD EXISTS OR WILL BE CREATED).



Principal Investigator: Niraj Desai, MD Application No.: IRB00237097

#### DOCUMENTATION OF PHYSICIAN/MID-LEVEL PROVIDER CONSENT

My signature below indicates that I have discussed the risks, benefits, and alternatives, answered any questions, and believe the participant is able to make an informed choice to join the study.

| Signature of Physician/Mid-Level Provider | (Print Name) | Date/Time |
|---|---|---|
| Signature of Participant | (Print Name) | Date/Time |
| Signature of Interpreter/Witness to Consent Procedures | (Print Name) | Date/Time |

NOTE: A COPY OF THE SIGNED, DATED CONSENT FORM MUST BE KEPT BY THE PRINCIPAL INVESTIGATOR AND A COPY MUST BE GIVEN TO THE PARTICIPANT. IF APPROPRIATE FOR THIS STUDY, A SCANNED COPY OF THE SIGNED CONSENT FORM SHOULD BE UPLOADED TO THE PARTICIPANT'S EPIC/EMR RECORD (UNLESS NO MEDICAL RECORD EXISTS OR WILL BE CREATED).